CLINICAL TRIAL: NCT03950648
Title: Spatial Cognitive Training for Chronic Vestibular Disorders
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: University of Pittsburgh (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Brooke Klatt, Postdoctoral Research Fellow, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19030436
Record Dates: First submitted 2019-05-11; First posted 2019-05-15 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Vestibular Abnormality; Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spatial Cognitive Training (Experimental): map reading and route-learning skills
  Interventions: Behavioral: Spatial Cognitive Training

INTERVENTIONS:
Behavioral: Spatial Cognitive Training — map reading and route-learning skills

SUMMARY:
In this study the investigators propose to apply cognitive training, which has been largely used in the realm of age-related cognitive decline, dementia, and Alzheimer's disease, in a novel clinical context to individuals with vestibular impairment. In prior work the investigators observed that individuals with vestibular loss have evidence of spatial cognitive impairment. The investigators plan to evaluate the preliminary efficacy and feasibility of a cognitive training program in a sample of participants with chronic vestibular impairment who display deficits in spatial ability. The cognitive training program will focus on visuospatial skills and will be used as an adjunct to traditional vestibular physical therapy (VPT).

DETAILED DESCRIPTION:
Patients with chronic vestibular dysfunction with report symptoms of spatial cognitive impairment will be offered cognitive training. The intervention will consist of a well-validated cognitive training protocol that specifically targets spatial navigation skills. The protocol was developed by Willis et al. for the Adult Development and Enrichment Trial (ADEPT) trial, which trains map reading and route-learning skills through mental rotation training tasks over the course of 5 weeks. Patients will be assessed by study staff pre-intervention, immediately post-intervention and at 3 months post-intervention using spatial cognitive outcomes, quality of life measures, and gait and balance outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic vestibular disorder (>6months & diagnosis from laboratory testing by neuro-otologist)

Exclusion Criteria:

* Participants with dementia, or with blindness or deafness who cannot participate in cognitive training procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Dizziness Handicap Inventory | Baseline vs immediately post-training
  Subjective 25-item questionnaire measuring Quality of Life and disability on a scale from 0-100
Change from immediate post-training to 3-months post-training in Dizziness Handicap Inventory | Immediately post-training to 3 months post-training
  Subjective 25-item questionnaire measuring Quality of Life and disability on a scale from 0-100
Change from baseline in Dynamic Gait Index | Baseline vs immediately post-training
  Balance challenges during 8 different gait tasks (head turns, speed changes, over/around obstacles) with total score out of 24 points.
Change from immediate post-training to 3-months post-training in Dynamic Gait Index | Immediately post-training to 3 months post-training
  Balance challenges during 8 different gait tasks (head turns, speed changes, over/around obstacles) with total score out of 24 points.
Change from baseline in Four Square Step Test | Baseline vs immediately post-training
  Assesses dynamic balance, spatial, & sequencing skills while stepping forward/back/sideways over a low obstacle (measured in seconds)
Change from immediate post-training to 3-months post-training in Four Square Step Test | Immediately post-training to 3 months post-training
  Assesses dynamic balance, spatial, & sequencing skills while stepping forward/back/sideways over a low obstacle (measured in seconds)

SECONDARY OUTCOMES:
Change from baseline in Money Road Map Test | Baseline vs immediately post-training
  Assessment of egocentric mental rotation in space by recording total number of errors in right-left discrimination mental rotation tasks.
Change from immediate post-training to 3-months post-training in Money Road Map Test | Immediately post-training to 3 months post-training
  Assessment of egocentric mental rotation in space by recording total number of errors in right-left discrimination mental rotation tasks.
Change from baseline in Benton Visual Retention Test | Baseline vs immediately post-training
  visual perception and visual memory assessment by asking participant to reproduce 10 designs following a 10-second exposure and scored 0-10 based on correct drawing reconstruction.
Change from immediate post-training to 3-months post-training in Benton Visual Retention Test | Immediately post-training to 3 months post-training
  visual perception and visual memory assessment by asking participant to reproduce 10 designs following a 10-second exposure and scored 0-10 based on correct drawing reconstruction.
Change from baseline in modified Clinical Test of Sensory Organization and Balance | Baseline vs immediately post-training
  Static standing balance during 4 conditions where sensory inputs are altered (eyes open/eyes closed on firm/foam surface) and each condition is timed for max of 30 seconds.
Change from immediate post-training to 3-months post-training in modified Clinical Test of Sensory Organization and Balance | Immediately post-training to 3 months post-training
  Static standing balance during 4 conditions where sensory inputs are altered (eyes open/eyes closed on firm/foam surface) and each condition is timed for max of 30 seconds.
Change from baseline in Activities-specific Balance Confidence Scale | Baseline vs immediately post-training
  Subjective questionnaire that determines confidence during daily tasks (scores range 0-100%)
Change from immediate post-training to 3-months post-training in Activities-specific Balance Confidence Scale | Immediately post-training to 3 months post-training
  Subjective questionnaire that determines confidence during daily tasks (scores range 0-100%)
Change from baseline in Santa Barbara Sense of Direction Scale | Baseline vs immediately post-training
  15 question related to subjective sense of direction adeptness (ranging 1-7 for each item); cumulative score is divided by number of responses answered to yield a 1-7 total score.
Change from immediate post-training to 3-months post-training in Santa Barbara Sense of Direction Scale | Immediately post-training to 3 months post-training
  15 question related to subjective sense of direction adeptness (ranging 1-7 for each item); cumulative score is divided by number of responses answered to yield a 1-7 total score.

CONTACTS AND LOCATIONS:
Overall Officials: Brooke Klatt, PhD, PT, Principal Investigator — University of Pittsburgh

IPD SHARING:
Plan to Share IPD: Yes
dissemination of study findings in manuscript publication in scientific journal
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 1 year